CLINICAL TRIAL: NCT04540653
Title: Immunogenicity of the Hepatitis B Vaccine in Individuals 50 Years Old or More: Randomized Clinical Trial
Brief Title: Immunogenicity of the Hepatitis B Vaccine
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidade Federal de Goias (Other)
Responsible Party: Principal Investigator, Karlla Antonieta Amorim Caetano, Clinical Professor, Universidade Federal de Goias
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PI02102-2017
Record Dates: First submitted 2020-08-31; First posted 2020-09-07 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Vaccine Response Impaired; Hepatitis B; Aging
Keywords: Vaccine Response Impaired; Hepatitis B; Aging
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Intervention Model Description: The intervention group (Reinforced Intervention Scheme - EIR) indicates 3 doses of 40 μg (2 mL) of hepatitis B vaccine, in months 0, 1 and 6, while the comparison group (Conventional Comparison Scheme - ECC) completes 3 doses of 20 μg (1 mL) of the vaccine, in months 0, 1 and 6. To evaluate the kinetics of the hepatitis B vaccine, after each dose administered, about 30 to 60 days, 5 mL of blood was again collected from the participants for quantitative detection of anti-HBs, using the Microparticle Chemiluminescent Immunoassay (CMIA) method, according to the manufacturer's instructions.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard vaccination schedule (Other): To evaluate the immunogenicity of the monovalent hepatitis B vaccine, expressed in Hansenula polymorpha, aged ≥50 years old, using a standard vaccination schedule (three doses of 20 μg, in months 0, 1, 6).
  Interventions: Biological: Standard vaccination schedule
- Reinforced vaccination schedule (Experimental): To evaluate the immunogenicity of the monovalent hepatitis B vaccine, expressed in Hansenula polymorpha, in individuals aged ≥50 years, using a reinforced vaccination schedule (three doses of 40 μg, in months 0, 1, 6).
  Interventions: Biological: Reinforced vaccination schedule

INTERVENTIONS:
Biological: Standard vaccination schedule — Administer a standard vaccination schedule (three doses of 20 μg of the hepatitis B vaccine, in months 0, 1, 6) at an age of ≥50 years and evaluate a production kinetics after each dose administered in the period of about 30 to 60 days.
  Arms: Standard vaccination schedule
Biological: Reinforced vaccination schedule — Administer an enhanced vaccination schedule (three doses of 40 μg of the hepatitis B vaccine, in months 0, 1, 6) in individuals aged ≥50 years and assess the kinetics of antibody production after each dose administered in the period of approximately 30 to 60 days.
  Arms: Reinforced vaccination schedule

SUMMARY:
More than five decades have passed since the identification of the etiologic agent of hepatitis B and yet this infection is a challenge for public health worldwide. The development and availability of the first hepatitis B vaccines, still in the 1980s, was a milestone for the prevention of the hepatitis B virus, and currently known as the gold standard strategy for the elimination of this infectious disease.

In several countries, the introduction of the immunobiological occurred gradually, by age groups and risk groups, and in general, started with newborns and children. This universal immunization strategy has contributed to reducing the incidence and changing the epidemiological profile of HBV worldwide. At the beginning of the 21st century, it was already possible to shift the epidemiological curve of the infection to parasitize with 50 years or more. On the other hand, despite vaccination against hepatitis B being the most assertive tool for the prevention of HBV, the low performance of the vaccine in older groups remains a challenge for public health and the object of this study. To our knowledge, there are no data showing the efficacy of doses of enhanced hepatitis B vaccines for older adults, and the purpose of this study is to investigate and compare the immunogenicity of the hepatitis B vaccine in adult adults aged 50 years and over, using conventional doses (20μg) versus (vs) booster doses.

DETAILED DESCRIPTION:
More than five decades have passed since the identification of the etiologic agent of hepatitis B and yet this infection is a challenge for public health worldwide. The development and availability of the first hepatitis B vaccines, still in the 1980s, was a milestone for the prevention of the hepatitis B virus, and currently known as the gold standard strategy for the elimination of this infectious disease.

In several countries, the introduction of the immunobiological occurred gradually, by age groups and risk groups, and in general, started with newborns and children. In Brazil, only in 2015, a free offer of the hepatitis B vaccine expanded a population aged 50 years or older. This universal immunization strategy has contributed to reducing the incidence and changing the epidemiological profile of HBV worldwide. At the beginning of the 21st century, it was already possible to shift the epidemiological curve of the infection to parasitize with 50 years or more.

Consider this scenario of vulnerability to HBV in older adults, it is important to highlight some aspects. The increase in life expectancy around the world is real data and must be evaluated. In addition, contemporary aging is accompanied by an increase and improvement in sexual performance, overcoming myths about "asexual old age" and outdated stereotypes about sexuality for an adult population in the middle and late stages. On the other hand, sexual risk behavior in older people being observed, including unprotected sexual intercourse, multiple sexual partnerships, sexual intercourse with a sex worker, among others. Studies have been increasing the high prevalence of Sexually Transmitted Infections, especially hepatitis B in the elderly.

Given this situation, hepatitis B vaccination is the most assertive tool for preventing HBV. However, even in countries that expand the offer of the vaccine to the entire population, poor performance of the hepatitis B vaccine in older groups remains a challenge for public health and is the object of this study.

A study conducted by Meeren and collaborators, characterized the relationship age vs. age. vaccine response to hepatitis B in immunocompetent adults. The protection index identified, considering all age groups, was 94.5%. However, there was a continuous reduction in seroprotection associated with age, ranging from 98.6% for young adults aged 20-24 years to 64.8% for the elderly (≥65 years). In addition, this study suggested that the aging of the immune system starts in adulthood and is intensified after 50-60 years of age.

In the United States, research conducted with competence aged ≥50 years, showed lower rates of seroconversion compared to younger people, with protection rates ranging from 68% to 82.2%. Another study carried out in this country, elucidated the risk of non-response to the anti-HBV vaccine in 63% for products ≥40 years old (p = 0.046).

Finally, in Brazil, an investigation conducted by Caetano et al. with settlers in Goiás, also illustrated a low responsiveness to the hepatitis B vaccine in the older population. In the age group aged 40-49 years, seroprotection was identified in only 61.9% of the participants, and for the age group aged 50-59 years the rate of seroresponse was even lower, only 55.9% protective titles of anti- HBs. Another study with this same population in Mato Grosso do Sul, showed an average age above 40 years for our non-responders.

Thus, the program that supplants this limitation is necessary, until the cohort of children immunized at birth from a late adulthood. The use of third generation vaccines for this population seems to be difficult to implement due to the high cost of this immunogen. In this way, more frequent or more concentrated doses of the second generation vaccine can be a safe alternative for the older population.

To our knowledge, there are no data showing the efficacy of doses of enhanced hepatitis B vaccines for older adults, and the purpose of this study is to investigate and compare the immunogenicity of the hepatitis B vaccine in adult adults aged 50 years and over, using conventional doses (20μg) versus (vs) booster doses.

ELIGIBILITY:
Inclusion Criteria:

* person is 50 years of age or older.

Exclusion Criteria:

* people with chronic renal failure, cancer and HIV / AIDS, using corticosteroids;
* people with a history of hepatitis B vaccination (vaccination record of hepatitis B vaccine doses or previous report of hepatitis B vaccination);
* people who are positive for anti-HBs and / or total anti-HBc serological markers.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2017-07-29 (Actual); Primary Completion 2020-07-03 (Actual); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
More than 90% of the appropriate intervention sample of associated anti-HBs (≥10mUI / mL) after three doses of hepatitis B vaccine | Success of the proposed procedure, defined by the development of isolated anti-HBs titers (≥10mUI / mL) after three reinforced doses (40μg) of the hepatitis B vaccine, in 30 to 60 days after the end of the vaccination schedule.
  Success of the proposed procedure, defined by the development of isolated anti-HBs titers (≥10mUI / mL) after three reinforced doses (40μg) of the hepatitis B vaccine, within 30 to 60 days after the end of the vaccination schedule.

SECONDARY OUTCOMES:
About 20-30% of the appropriate intervention sample of associated anti-HBs (≥10mUI / mL) after first dose of hepatitis B vaccine | Success of the proposed procedure, defined by the development of isolated anti-HBs titers (≥10mUI / mL) after one reinforced dose (40μg) of the hepatitis B vaccine, within 30 to 60 days after the end of the vaccination schedule.
  Success of the proposed procedure, defined by the development of isolated anti-HBs titers (≥10mUI / mL) after one reinforced dose (40μg) of the hepatitis B vaccine, within 30 to 60 days after the end of the vaccination schedule.
About 75-80% of the appropriate intervention sample of associated anti-HBs (≥10mUI / mL) after second dose of hepatitis B vaccine | Success of the proposed procedure, defined by the development of isolated anti-HBs titers (≥10mUI / mL) after two reinforced doses (40μg) of the hepatitis B vaccine, within 30 to 60 days after the end of the vaccination schedule.
  Success of the proposed procedure, defined by the development of isolated anti-HBs titers (≥10mUI / mL) after two reinforced doses (40μg) of the hepatitis B vaccine, within 30 to 60 days after the end of the vaccination schedule.

CONTACTS AND LOCATIONS:
Overall Officials: Karlla Caetano, PhD, Principal Investigator — Universidade Federal de Goiás
Locations (1):
- Karlla Antonieta Amorim Caetano, Goiânia, Goiás, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aguiar RB, Leal MCC, Marques APO, Torres KMS, Tavares MTDB. [Elderly people living with HIV - behavior and knowledge about sexuality: an integrative review]. Cien Saude Colet. 2020 Feb;25(2):575-584. doi: 10.1590/1413-81232020252.12052018. Epub 2018 Jun 27. Portuguese. PMID 32022197
- [Background] Bastos LM, Tolentino JMS, Frota MAO, Tomaz WC, Fialho MLS, Batista ACB, Teixeira AKM, Barbosa FCB. [Evaluation of the level of knowledge about Aids and syphilis among the elderly from a city in the interior of the state of Ceara, Brazil]. Cien Saude Colet. 2018 Aug;23(8):2495-2502. doi: 10.1590/1413-81232018238.10072016. Portuguese. PMID 30137119
- [Background] BLUMBERG BS, ALTER HJ, VISNICH S. A "NEW" ANTIGEN IN LEUKEMIA SERA. JAMA. 1965 Feb 15;191:541-6. doi: 10.1001/jama.1965.03080070025007. No abstract available. PMID 14239025
- [Background] Caetano KA, Del-Rios NH, Pinheiro RS, Bergamaschi FP, Carneiro MA, Teles SA. Low Immunogenicity of Recombinant Hepatitis B Vaccine Derived from Hansenula polymorpha in Adults Aged Over 40 Years. Am J Trop Med Hyg. 2017 Jan 11;96(1):118-121. doi: 10.4269/ajtmh.16-0475. Epub 2016 Oct 31. PMID 27799647
- [Background] Gerlich WH. Prophylactic vaccination against hepatitis B: achievements, challenges and perspectives. Med Microbiol Immunol. 2015 Feb;204(1):39-55. doi: 10.1007/s00430-014-0373-y. Epub 2014 Dec 19. PMID 25523195
- [Background] Gilbert CL, Klopfer SO, Martin JC, Schodel FP, Bhuyan PK. Safety and immunogenicity of a modified process hepatitis B vaccine in healthy adults >/=50 years. Hum Vaccin. 2011 Dec;7(12):1336-42. doi: 10.4161/hv.7.12.18333. Epub 2011 Dec 1. PMID 22185811
- [Background] Liu Z, Yang Q, Shi O, Ye W, Chen X, Zhang T. The epidemiology of hepatitis B and hepatitis C infections in China from 2004 to 2014: An observational population-based study. J Viral Hepat. 2018 Dec;25(12):1543-1554. doi: 10.1111/jvh.12938. Epub 2018 Jun 20. PMID 29851287
- [Background] Lyons A, Heywood W, Fileborn B, Minichiello V, Barrett C, Brown G, Hinchliff S, Malta S, Crameri P. The Sex, Age, and Me study: recruitment and sampling for a large mixed-methods study of sexual health and relationships in an older Australian population. Cult Health Sex. 2017 Sep;19(9):1038-1052. doi: 10.1080/13691058.2017.1288268. Epub 2017 Feb 21. PMID 28276921
- [Background] Van Der Meeren O, Crasta P, Cheuvart B, De Ridder M. Characterization of an age-response relationship to GSK's recombinant hepatitis B vaccine in healthy adults: An integrated analysis. Hum Vaccin Immunother. 2015;11(7):1726-9. doi: 10.1080/21645515.2015.1039758. PMID 25996260
- [Background] Minichiello V, Rahman S, Hawkes G, Pitts M. STI epidemiology in the global older population: emerging challenges. Perspect Public Health. 2012 Jul;132(4):178-81. doi: 10.1177/1757913912445688. PMID 22729008
- [Background] Monsell E, McLuskey J. Factors influencing STI transmission in middle-aged heterosexual individuals. Br J Nurs. 2016 Jun 23;25(12):676-80. doi: 10.12968/bjon.2016.25.12.676. PMID 27345071
- [Background] Rosenberg C, Bovin NV, Bram LV, Flyvbjerg E, Erlandsen M, Vorup-Jensen T, Petersen E. Age is an important determinant in humoral and T cell responses to immunization with hepatitis B surface antigen. Hum Vaccin Immunother. 2013 Jul;9(7):1466-76. doi: 10.4161/hv.24480. Epub 2013 Apr 9. PMID 23571167
- [Background] Sagnelli E, Stroffolini T, Sagnelli C, Morisco F, Coppola N, Smedile A, Pisaturo M, Colloredo G, Babudieri S, Licata A, Brancaccio G, Andriulli A, Almasio PL, Gaeta GB; EPACRON study group. Influence of universal HBV vaccination on chronic HBV infection in Italy: Results of a cross-sectional multicenter study. J Med Virol. 2017 Dec;89(12):2138-2143. doi: 10.1002/jmv.24873. Epub 2017 Aug 29. PMID 28608566
- [Background] Sharma R, Ahlm C, Ostergaard L, Dowell A, Tran C, Thomas S, Eymin C. Persistence of immunity in healthy adults aged >/= 50 years primed with a hepatitis B vaccine 3 years previously. Hum Vaccin Immunother. 2015;11(7):1709-16. doi: 10.1080/21645515.2015.1019187. PMID 25996838
- [Background] Szmuness W, Stevens CE, Harley EJ, Zang EA, Oleszko WR, William DC, Sadovsky R, Morrison JM, Kellner A. Hepatitis B vaccine: demonstration of efficacy in a controlled clinical trial in a high-risk population in the United States. N Engl J Med. 1980 Oct 9;303(15):833-41. doi: 10.1056/NEJM198010093031501. PMID 6997738
- [Background] Tran TQ, Grimes CZ, Lai D, Troisi CL, Hwang LY. Effect of age and frequency of injections on immune response to hepatitis B vaccination in drug users. Vaccine. 2012 Jan 5;30(2):342-9. doi: 10.1016/j.vaccine.2011.10.084. Epub 2011 Nov 8. PMID 22075088
- [Background] Vermeulen M, Swanevelder R, Chowdhury D, Ingram C, Reddy R, Bloch EM, Custer BS, Murphy EL; NHLBI Recipient Epidemiology and Donor evaluation Study-III (REDS-III) International Component. Use of Blood Donor Screening to Monitor Prevalence of HIV and Hepatitis B and C Viruses, South Africa. Emerg Infect Dis. 2017 Sep;23(9):1560-1563. doi: 10.3201/eid2309.161594. PMID 28820374
- See also: WHO; World Health Organization. Global Hepatitis Report 2017. Geneva: WHO; 2017. — https://www.who.int/hepatitis/publications/global-hepatitis-report2017/en/
- See also: United Nations; Department of Economic and Social Affairs, Population Division (2019). World Population Ageing 2019. New York: United Nations; 2019. — https://www.un.org/en/development/desa/population/publications/pdf/ageing/WorldPopulationAgeing2019-Highlights.pdf
- See also: Bergamaschi FPR. Epidemiologia da infecção pelo vírus da hepatite b em assentamento rural em Mato Grosso do Sul, Brasil Central [Tese]. Goiânia-GO: Universidade Federal de Goiás; 2013. 95p — https://repositorio.bc.ufg.br/tede/handle/tede/3785